# COMIRB Protocol

COLORADO MULTIPLE INSTITUTIONAL REVIEW BOARD

CAMPUS BOX F-490 TELEPHONE: 303-724-1055 Fax: 303-724-0990

**Protocol #: 20-1866** 

Project Title: Understanding Affective Processing of Scientific Evidence to Promote Informed

Choice for Breast Cancer Screening

Principal Investigator: Laura Scherer, PhD

**Version Date: 5.10.2021** 

## I. Hypotheses and Specific Aims:

Cancer screening for the right patients at the right level of cancer risk can save lives. However, over the last several years most expert groups have de-intensified many screening recommendations as a result of emerging evidence of net harms for certain populations. Newer recommendations for mammography screening highlight a tailored approach based on age and risk and comorbidities, aiming to minimize harms and target women who could benefit the most.<sup>1</sup> Although there is still widespread disagreement about when and how frequently certain populations of women should receive breast screening, one point of agreement is that women should make an informed choice with their doctor about when to start, when to stop, and how frequently to screen.<sup>2–</sup>

However, the change in emphasis from uniformly promoting mammography to promoting informed choice constitutes a medical reversal in the sense that this new message is very different from past messages and people's expectations. The result is a delicate situation in which there is need to convey the evidence to women, but also a need to do it in a way that maintains credibility and trust despite this reversal. Research suggests that many women react negatively to mammography evidence, responding with Reactance (e.g., "this is trying to manipulate me", "this is trying to ration healthcare"), self-Exemption (e.g., "this doesn't apply to me"), Disbelief (e.g., "you can't believe all the research"), or Source derogation (e.g., "I don't trust this source"), 6,8,9 which we refer to together as REDS. These responses reflect different ways of rejecting of the evidence, stand in the way of informed choice, and could lead to distrust in future screening health messages.

AIM 1: Identify the prevalence and predictors of REDS in reaction to evidence about mammography benefits and harms, and consequences for decision-making and trust. Research has not yet systematically identified the proportion of women who respond negatively (vs. positively) to mammography evidence, or attempted to explain these responses by examining theory-driven predictors. We will develop and conduct a probability-based nationally representative survey in which we communicate mammography evidence using the current best practices in risk communication, and identify theory-driven predictors of REDS responses, and identify consequences of these responses for decision-making and trust.

#### II. Background and Significance:

A1. Screening recommendations have changed considerably over recent years.

Breast cancer is the second leading cause of cancer death among women in the U.S., and early detection can result in a cure before it spreads. For many years mammography was strongly promoted, with the aim of maximizing screening uptake. 10–12 However, mammography guidelines have changed considerably as a result of accumulating evidence showing that screening has less benefit for some populations of women, and can cause harm. 13–15 Harms include false positive results requiring follow-up tests and biopsies, and overdiagnosis—the diagnosis of asymptomatic cancer that will not cause symptoms or harm in a person's lifetime—and resultant overtreatment. 16–18 Although routine mammography is still strongly recommended for women in specific age ranges

and with certain risk factors, many expert groups, including the United States Preventive Services Task Force (USPSTF) and the American Cancer Society (ACS), have de-intensified screening recommendations and expanded the role of informed choice.<sup>2,4</sup> Most guidelines now emphasize that women should receive balanced information about the benefits and harms of mammography so that they can engaged in shared decision making (SDM) and make an informed choice with their doctor about when to start, when to stop, and how frequently to screen.<sup>19</sup>

A2. A balanced presentation of both screening benefits and harms is very different from previous unequivocal recommendations to screen, and can strongly contradict women's preexisting beliefs. Controversies about breast cancer screening continues to receive attention in the news media but many women are still unaware of the evidence.<sup>20,21</sup> Most women greatly overestimate their lifetime breast cancer risk,22 and overestimate their risk even after they have been counseled on their objective risk.<sup>23</sup> A recent systematic review found that in 8 of 9 studies reviewed, a majority (i.e. >50%) of women overestimated the benefit of mammography.<sup>24</sup> Most people (women and men) have little or no prior knowledge of harm from overdiagnosis, which is a counterintuitive concept that contradicts common beliefs about how cancer grows and spreads.<sup>5,25–28</sup> In a 2016 survey, only 16% of women were aware of overdiagnosis as a harm of mammography.6 Screening is rarely discussed in clinical encounters in a balanced way; for example, in one survey only 19% of women reported that their provider had discussed the harms of screening in addition to the benefits.<sup>29</sup> The public is also very enthusiastic about cancer screening. 10,30,31 For example, in a recent study we found that 43% of women and men expressed a desire for breast/prostate cancer screening even if it would not reduce the chance of cancer death or extend the length of life.30

A3. Mammography evidence and revised quidelines can be emotionally charged. "It feels like just when it became okay to talk about breasts and screening, and we convinced insurance to pay for it, and we started getting it to low income women, now we're told that it's maybe not that great and it should be a choice. How are we supposed to believe that?" (personal communication with PI Scherer). Given that many women overestimate their breast cancer risk and the benefits of screening, are unaware of the harms of screening, and are very enthusiastic about screening, it should come as no surprise that mammography evidence and the recommendation for informed choice can elicit negative reactions. Qualitative research has shown that some women are suspicious and resistant to screening evidence, particularly the notion of overdiagnosis.<sup>32</sup> In a 2016 U.S. survey less than 1-in-4 women thought both overdiagnosis and overtreatment were "believable". 6 The notion of risk-based screening—that is, creating a screening plan tailored to a woman's objective cancer risk—is concerning for some women, and can raise suspicions of healthcare rationing.<sup>20</sup> In a recent study, women rated a leaflet that described the balance of benefits and harms as less helpful than one that promoted only the benefits, which the authors interpreted as potentially indicating a reluctance to accept information about harms.<sup>33</sup> In recent focus groups involving 42 U.S. adults, participants placed enormous value on cancer screening and expressed hostility toward guidelines suggesting doing less screening.<sup>34</sup> Recently we conducted 16 patient interviews in anticipation of this proposal in which we showed women a breast cancer screening decision support tool35 and asked how they felt about the benefits and harms presented. Here is how one woman responded to the idea of harm from overdiagnosis: "I think this might give people a false sense of security. Like it's giving them permission to not do screening. So I don't think that this is reassuring, and I don't think it accurately represents the actual risk. This whole thing kinda makes me mad. I find it very frustrating because it, it feels like...it feels like propaganda."

Altogether, the weight of the evidence suggests that communicating mammography screening evidence can elicit negative reactions. The types of negative reactions that we are particularly concerned about include **Reactance** (i.e. perceived manipulation or influence, e.g. "this is trying to ration healthcare"), **self-Exemption** (e.g., "this doesn't apply to me"), **Disbelief** (e.g., "you can't believe all the research anyway"), and **Source derogation** (e.g., "I don't trust this source"), which we shorten to **REDS**. "These responses are sometimes referred to collectively as "defensive coping", although we prefer "REDS" to refer directly to the four types of responses. To date, no research has examined REDS systematically to assess their prevalence and causes in the context of communicating mammography screening evidence. And even though many women

react negatively to screening information, many women also want to be informed and be able to make a choice.<sup>37</sup> The result is a delicate situation in which there is need to convey the evidence to women, but also a need to do it in a way that maintains credibility and trust.

## III. Preliminary Studies/Progress Report:

### IV. Research Methods

## A. Outcome Measure(s):

The primary outcome measures in this survey are REDS responses and screening intentions. See Table 1 below for all survey measures. <sup>35,55,56,61,66,72,96–99</sup>

| | Measure description | Source |
|---|---|---|
| Primary<br>DVs | REDS responses | See appendix |
| | Screening intentions | Schapira et al. 2019 |
| Secondary<br>DVs | Change in trust in provider and healthcare system, pre vs. post BCS-DA | Egede et al. 2008 |
| | Positive responses, e.g. appreciation of information | Ad hoc |
| | Change in screening knowledge, pre vs. post BCS-DA | Schapira et al. 2019 |
| IVs:<br>primary | Breast cancer risk perceptions: affective, deliberative, experiential | Ferrer et al. 2016 |
| | Perception of net screening benefit (benefits minus harms) at pre-test | Scherer et al., 2018 |
| | Objective breast cancer risk | Schapira et al. 2019 |
| | Cognitive responses to information | See appendix |
| | Medical Maximizing-Minimizing orientation | Scherer et al., 2016 |
| | Perceived norms | Hersch et al., 2015 |
| | Past screening experience | Petrova et al., 2015 |
| Secondary<br>IVs and<br>control<br>variables | Perceived barriers to screening | Hyman & Baker 1992 |
| | Friends/family experience with breast cancer | Petrova et al., 2015 |
| | Subjective numeracy | Fagerlin et al., 2007 |
| | Health literacy | Chew et al., 2008 |
| | Demographics | Standard questions |

Table 1. Aim 1 measures.

### B. Description of Population to be Enrolled:

## Inclusion:

- Female
- Between 39-49 years of age
- No history of breast cancer
- No known BRCA1/2 mutation

### Exclusion:

- Non-English or Spanish Speaking
- Persons unable to provide informed consent (e.g. severe dementia or cognitive disability or illiterate)
- History of breast cancer
- Known BRCA1/2 mutation

Pilot Survey: We will pilot test questions to measure REDS and cognitive reactions to assess item variability, internal consistency, and reduce the total number of items. We will recruit 700 women through Dynata. Dynata manages an online participant panel of millions of adults across the United States. Participants who are part of Dynata's panel have agreed to participate in surveys in exchange entry into lotteries for small cash prizes.

Pilot Interviews: We will recruit up to 15 women from Carmen Lewis's Internal Medicine clinic at UCHealth. These interviews will focus on assessing overall knowledge and understanding of the information presented in the decision aid. Participants will receive a \$25 gift card for participating in the interview.

Nationally Representative Survey: We will recruit 700 women age 40-49 through Ipsos Public Affairs. Ipsos manages an online participant panel allowing population inferences using probability sampling methods and providing Internet access to households that do not have it.

Nationally Representative Interviews: We will recruit up to 40 women from the Ipsos survey who agreed to be contact for a follow-up phone interview. We will specifically recruit women who expressed negative reactions to mammography evidence, so that we can assess how to improve the BCS-DA using insights from those who were negatively affected. We will attempt to recruit at least 25% non-White participants for these interviews.

## C. Study Design and Research Methods

 Knowledge of Cancer risk, screening benefit & harm Perception of screening benefit and harm • Trust in healthcare and physicians Premeasures · Screening intentions in next 12 months Perceived social norms about screening • Risk calculator questions • Risk perceptions: Affective Risk calculator Deliberative results Experiential REDS responses REDS responses Harm evidence: Cognitive responses False positives REDS responses Harm evidence: Over diagnosis Overall REDS responses Overall cognitive responses Final evaluation • Overall positive responses, e.g. appreciation of of evidence information Knowledge of cancer risk, screening benefit & harm • Perception of screening benefit and harm • Trust in healthcare and physicians measures • Screening intentions in next 12 months • Medical Maximizer-Minimizer Scale Subjective numeracy Health Literacy Individual • Past screening experiences difference • Friends & family cancer experiences measure Perceived barriers • Standard demographics

The survey flow is displayed in the figure below and will unfold as follows: First. women will be asked premeasure questions displayed in the figure below. Second, women will learn their objective cancer risk estimate, and will report their affective, deliberative and experiential risk perceptions. <sup>56</sup> Third, women will react separately to the three distinct components of mammography evidence (benefits, false positives, overdiagnosis). The purpose of assessing reactions to each component of the evidence is to identify how positively or negatively each part is received. We anticipate that overdiagnosis may be received most negatively. Measured reactions will include REDS responses, and cognitive reactions as previously described (i.e. whether the information is compatible or not with other knowledge). Finally, after all of the information has been presented, women will provide overall reactions to

the evidence using the same measures. Next women will report overall positive responses, e.g., the extent to which they appreciated receiving the information, felt empowered by it, and

want to talk to their provider about it. Lastly, women will repeat some of the pre-measures (e.g. knowledge, trust) and report demographics and individual differences.

Pilot Survey: Recruitment and survey distribution with be done by Dynata. All data will be collected electronically using Qualtrics.

Nationally Representation Survey: Recruitment and survey distribution with be done by Ipsos. All data will be collected electronically using Qualtrics.

All Interviews: Patients will be invited to schedule a phone call for the interview (using a regular phone or using Zoom), and audio will be recorded and transcribed.

## D. Description, Risks and Justification of Procedures and Data Collection Tools:

Benefit from participating in the research cannot be claimed. Women will learn about mammography benefit and harm, which may lead to more informed screening decisions. Learning how to help communicate more effectively about counterintuitive and surprising medical evidence is an area in great need of attention. The intervention is designed to improve communication and decision quality and enhance the overall decision making. Given that the risks are minimal and the benefits great (to both patients, clinicians, and society as a whole) we believe that the benefits of the proposed project outweigh any risks.

#### E. Potential Scientific Problems:

The length of the survey may be an issue since we are recruiting through Ipsos.

There is a possibility that not a sufficient amount of subjects with voluntarily self-identify for the follow-up interviews.

### F. Data Analysis Plan:

Pilot Survey: We will check the variability of each questionnaire item to assess suitability for exploratory factor analysis. Exploratory factor analysis will be used to identify the factor structure of the REDS items. Items that do not load onto any factor will be dropped. Reliability of the remaining items

Nationally Representative Survey: Summary statistics will estimate the prevalence of REDS to each part of the BCS-DA. Simple within-subjects tests (e.g. ANOVA) will compare REDS in response to screening benefits, false positives, and overdiagnosis.

All Interviews: We will conduct exploratory content analysis of these qualitative interviews using the analytic program Dedoose to extract themes in patients' reactions to the presented information.

## Safety Oversight:

The principal investigator will be responsible for the conduct of this study, overseeing participant safety, executing the data and safety monitoring (DSM) plan, and complying with all reporting requirements to local and federal authorities. This oversight will be accomplished through additional oversight from the Data and Safety Monitoring Committee (DSMC) at the University of Colorado Cancer Center (CU Cancer Center). The DSMC is responsible for ensuring data quality and study participant safety for all trials at the CU Cancer Center. A summary of the DSMC's relevant activities is as follows:

· Conduct of internal audits

- Has the authority to suspend studies for safety or conduct issues
- May submit recommendations for corrective actions to the CU Cancer Center's Executive Committee

Study audits conducted by the DSMC will consist of a review of the regulatory documents, consent forms, and source data verification. Documentation of the audit conducted by the DSMC will then need to be submitted to the IRB of record at the time of the IRB's continuing review of this trial (if applicable).

## G. Summarize Knowledge to be Gained:

Our preliminary data suggest that there are important problems with current approaches to communicating screening evidence. The proposed studies are designed to generate knowledge that will lead to improved communication strategies and real-world improvements in informed patient choice. Because virtually little work has systematically studied this issue, a deeper understanding of how women respond to screening evidence will have widespread clinical applicability.

### H. References:

- Squiers, L. B. et al. The Public's Response to the U.S. Preventive Services Task Force's 2009 Recommendations on Mammography Screening. Am. J. Prev. Med. 40, 497–504 (2011).
- 2. Oeffinger, K. C. *et al.* Breast Cancer Screening for Women at Average Risk: 2015 Guideline Update From the American Cancer Society. *JAMA* **314**, 1599 (2015).
- 3. Autier, P. & Boniol, M. Mammography screening: A major issue in medicine. *Eur. J. Cancer* **90**, 34–62 (2018).
- 4. U.S. Preventive Services Task Force. Final Recommendation Statement: Breast Cancer: Screening. (2016).
- 5. McCaffery, K. J. *et al.* Walking the tightrope: communicating overdiagnosis in modern healthcare. *BMJ* i348 (2016) doi:10.1136/bmj.i348.
- 6. Nagler, R. H., Franklin Fowler, E. & Gollust, S. E. Women's Awareness of and Responses to Messages About Breast Cancer Overdiagnosis and Overtreatment: Results From a 2016 National Survey. *Med. Care* **55**, 879–885 (2017).
- 7. Squiers, L. B. *et al.* Prostate-specific antigen testing: men's responses to 2012 recommendation against screening. *Am. J. Prev. Med.* **45**, 182–189 (2013).
- 8. Witte, K. Putting the fear back into fear appeals: The extended parallel process model. *Commun. Monogr.* **59**, 329–349 (1992).
- 9. Dillard, J. P. & Shen, L. On the Nature of Reactance and its Role in Persuasive Health Communication. *Commun. Monogr.* **72**, 144–168 (2005).
- 10. Schwartz, L. M., Woloshin, S., Fowler Jr, F. J. & Welch, H. G. Enthusiasm for cancer screening in the United States. *Jama* **291**, 71–78 (2004).
- 11. Mazor, K. M. *et al.* Media Messages About Cancer: What Do People Understand? *J. Health Commun.* **15**, 126–145 (2010).
- 12. Wang, A. T. *et al.* Impact of the 2009 US Preventive Services Task Force guidelines on screening mammography rates on women in their 40s. *PloS One* **9**, e91399 (2014).
- 13. US Preventive Services Task Force *et al.* Screening for Prostate Cancer: US Preventive Services Task Force Recommendation Statement. *JAMA* **319**, 1901 (2018).
- 14. Barry, M. J. Screening for Prostate Cancer The Controversy That Refuses to Die. *N. Engl. J. Med.* **360**, 1351–1354 (2009).
- 15. Allen, J. D. *et al.* Women's responses to changes in U.S. preventive task force's mammography screening guidelines: results of focus groups with ethnically diverse women. *BMC Public Health* **13**, (2013).
- 16. Carter, S. M. *et al.* The challenge of overdiagnosis begins with its definition. *BMJ* **350**, h869–h869 (2015).

- 17. Marcus, P. M., Prorok, P. C., Miller, A. B., DeVoto, E. J. & Kramer, B. S. Conceptualizing Overdiagnosis in Cancer Screening. *JNCI J. Natl. Cancer Inst.* **107**, djv014–djv014 (2015).
- 18. Welch, H. G. & others. Overdiagnosis and mammography screening. Bmj 339, (2009).
- 19. Spatz, E. S., Krumholz, H. M. & Moulton, B. W. Prime Time for Shared Decision Making. *JAMA* **317**, 1309 (2017).
- 20. He, X. et al. How Do Women View Risk-Based Mammography Screening? A Qualitative Study. J. Gen. Intern. Med. 33, 1905–1912 (2018).
- 21. Nagler, R. H., Fowler, E. F., Marino, N. M., Mentzer, K. M. & Gollust, S. E. The Evolution of Mammography Controversy in the News Media: A Content Analysis of Four Publicized Screening Recommendations, 2009 to 2016. *Womens Health Issues* **29**, 87–95 (2019).
- 22. Hoffman, R. M. *et al.* Knowledge and values for cancer screening decisions: Results from a national survey. *Patient Educ. Couns.* **99**, 624–630 (2016).
- 23. Lerman, C. *et al.* Effects of individualized breast cancer risk counseling: a randomized trial. *JNCI J. Natl. Cancer Inst.* **87**, 286–292 (1995).
- Hoffmann, T. C. & Del Mar, C. Patients' Expectations of the Benefits and Harms of Treatments, Screening, and Tests: A Systematic Review. *JAMA Intern. Med.* 175, 274 (2015).
- 25. Yu, J., Nagler, R. H., Fowler, E. F., Kerlikowske, K. & Gollust, S. E. Women's Awareness and Perceived Importance of the Harms and Benefits of Mammography Screening: Results From a 2016 National Survey. *JAMA Intern. Med.* (2017) doi:10.1001/jamainternmed.2017.2247.
- 26. Roberts, M. C. *et al.* Lay Beliefs About the Accuracy and Value of Cancer Screening. *Am. J. Prev. Med.* **54**, 699–703 (2018).
- 27. Hersch, J. et al. Women's views on overdiagnosis in breast cancer screening: a qualitative study. *BMJ* **346**, (2013).
- Sutkowi-Hemstreet, A. et al. Adult Patients' Perspectives on the Benefits and Harms of Overused Screening Tests: a Qualitative Study. J. Gen. Intern. Med. 30, 1618–1626 (2015).
- 29. Hoffman, R. M. *et al.* Decision-Making Processes for Breast, Colorectal, and Prostate Cancer Screening: The DECISIONS Survey. *Med. Decis. Making* **30**, 53S-64S (2010).
- 30. Scherer, L. D., Valentine, K., Patel, N. & Baker, S. G. A bias for action in cancer screening? *J. Exp. Psychol. Appl.* (in press).
- 31. Waller, J., Osborne, K. & Wardle, J. Enthusiasm for cancer screening in Great Britain: a general population survey. *Br. J. Cancer* **112**, 562–566 (2015).
- 32. Pappadis, M. R. *et al.* Perceptions of overdetection of breast cancer among women 70 years of age and older in the USA: a mixed-methods analysis. *BMJ Open* **8**, e022138 (2018)
- 33. Pérez-Lacasta, M. J. *et al.* Effect of information about the benefits and harms of mammography on women's decision making: The InforMa randomised controlled trial. *PLOS ONE* **14**, e0214057 (2019).
- 34. Schleifer, D. & Rothman, D. J. "The Ultimate Decision Is Yours": Exploring Patients' Attitudes about the Overuse of Medical Interventions. *PLoS ONE* **7**, e52552 (2012).
- 35. Hersch, J. *et al.* Use of a decision aid including information on overdetection to support informed choice about breast cancer screening: a randomised controlled trial. *The Lancet* **385**, 1642–1652 (2015).
- 36. McQueen, A., Vernon, S. W. & Swank, P. R. Construct definition and scale development for defensive information processing: An application to colorectal cancer screening. *Health Psychol.* **32**, 190–202 (2013).
- 37. Abelson, J., Tripp, L. & Sussman, J. 'I just want to be able to make a choice': Results from citizen deliberations about mammography screening in Ontario, Canada. *Health Policy* **122**, 1364–1371 (2018).
- 38. Lewandowsky, S., Ecker, U. K. H. & Cook, J. Beyond Misinformation: Understanding and Coping with the "Post-Truth" Era. *J. Appl. Res. Mem. Cogn.* **6**, 353–369 (2017).
- 39. Chou, W.-Y. S., Oh, A. & Klein, W. M. P. Addressing Health-Related Misinformation on Social Media. *JAMA* **320**, 2417–2418 (2018).

- 40. Navar, A. M. Fear-Based Medical Misinformation and Disease Prevention: From Vaccines to Statins. *JAMA Cardiol.* (2019) doi:10.1001/jamacardio.2019.1972.
- 41. Morgan, D. J., Dhruva, S. S., Coon, E. R., Wright, S. M. & Korenstein, D. 2018 Update on Medical Overuse. *JAMA Intern. Med.* (2018) doi:10.1001/jamainternmed.2018.5748.
- 42. Morgan, D. J., Dhruva, S. S., Coon, E. R., Wright, S. M. & Korenstein, D. 2017 Update on Medical Overuse: A Systematic Review. *JAMA Intern. Med.* 178, 110–115 (2018).
- 43. Cassel, C. K. & Guest, J. A. Choosing Wisely Helping Physicians and Patients Make Smart Decisions About Their Care. *JAMA J. Am. Med. Assoc.* **307**, 1801–1802 (2012).
- 44. Berwick, D. M. Avoiding overuse—the next quality frontier. *The Lancet* **390**, 102–104 (2017).
- 45. Brownlee, S. *et al.* Evidence for overuse of medical services around the world. *The Lancet* **390**, 156–168 (2017).
- 46. Saving Thyroids Overtreatment of Small Papillary Cancers | NEJM. https://www.nejm.org/doi/full/10.1056/NEJMp1804426.
- 47. Al-Lamee, R. *et al.* Percutaneous coronary intervention in stable angina (ORBITA): a double-blind, randomised controlled trial. *The Lancet* **391**, 31–40 (2018).
- 48. Druckman, J. N. & McGrath, M. C. The evidence for motivated reasoning in climate change preference formation. *Nat. Clim. Change* 1 (2019) doi:10.1038/s41558-018-0360-1.
- 49. McKenzie, C. R. M. The accuracy of intuitive judgment strategies: Covariation assessment and Bayesian inference. *Cognit. Psychol.* **26**, 209–209 (1994).
- 50. Piaget, J. The role of action in the development of thinking. in *Knowledge and development* 17–42 (Springer, 1977).
- 51. Johnson-Laird, P. N. Mental models of meaning. (1981).
- 52. Benyamini, Y. & Karademas, E. C. Introduction to the special issue on the common sense model of self-regulation. *Health Psychol. Rev.* **13**, 373–377 (2019).
- 53. Leventhal, H. Findings and theory in the study of fear communications. in *Advances in experimental social psychology* vol. 5 119–186 (Elsevier, 1970).
- 54. Janz, N. K. & Becker, M. H. The health belief model: A decade later. *Health Educ. Behav.* **11**, 1–47 (1984).
- 55. Hyman, R. B. & Baker, S. Construction of the Hyman-Baker mammography questionnaire, a measure of health belief model variables. *Psychol. Rep.* **71**, 1203–1215 (1992).
- 56. Ferrer, R. A., Klein, W. M. P., Persoskie, A., Avishai-Yitshak, A. & Sheeran, P. The Tripartite Model of Risk Perception (TRIRISK): Distinguishing Deliberative, Affective, and Experiential Components of Perceived Risk. *Ann. Behav. Med.* **50**, 653–663 (2016).
- 57. Slovic, P., Finucane, M. L., Peters, E. & MacGregor, D. G. Risk as analysis and risk as feelings: Some thoughts about affect, reason, risk, and rationality. *Risk Anal.* **24**, 311–322 (2004).
- 58. Festinger, L. A theory of cognitive dissonance. (Evanston: Row, Peterson, 1957).
- 59. Stiggelbout, A. *et al.* 87 Women's acceptance of overdetection in breast cancer screening: can we assess harm-benefit trade-offs? *BMJ Evid.-Based Med.* **23**, A41–A41 (2018).
- 60. Ajzen, I. The theory of planned behavior. *Organ. Behav. Hum. Decis. Process.* **50**, 179–211 (1991).
- 61. Scherer, L. D. *et al.* Development of the Medical Maximizer-Minimizer Scale. *Health Psychol.* **35**, 1276–1287 (2016).
- 62. Campbell, T., O'Brien, E., Van Boven, L., Schwarz, N. & Ubel, P. Too much experience: A desensitization bias in emotional perspective taking. *J. Pers. Soc. Psychol.* **106**, 272 (2014).
- 63. Wilson, T. D. & Gilbert, D. T. Explaining Away: A Model of Affective Adaptation. *Perspect. Psychol. Sci.* **3**, 370–386 (2008).
- 64. Pearlman, D. N. *et al.* Why do women's attitudes toward mammography change over time? Implications for physician-patient communication. *Cancer Epidemiol. Prev. Biomark.* **6**, 451–457 (1997).
- 65. Scherer, L. D. *et al.* Belief in numbers: When and why women disbelieve tailored breast cancer risk statistics. *Patient Educ. Couns.* **92**, 253–259 (2013).

- 66. Scherer, L. D. *et al.* The role of the affect heuristic and cancer anxiety in responding to negative information about medical tests. *Psychol. Health* **33**, 292–312 (2018).
- 67. Scherer, L. D. *et al.* Medical Maximizing-Minimizing Preferences Predict Responses to Information about Prostate Specific Antigen Screening. *Med. Decis. Making* (in press).
- 68. Schapira, M. M. *et al.* A framework for health numeracy: how patients use quantitative skills in health care. *J. Health Commun.* **13**. 501–517 (2008).
- 69. Schapira, M. M. *et al.* The relationship of health numeracy to cancer screening. *J. Cancer Educ.* **26**, 103–110 (2011).
- 70. Schapira, M. M. *et al.* The numeracy understanding in medicine instrument: a measure of health numeracy developed using item response theory. *Med. Decis. Making* **32**, 851–865 (2012).
- 71. Elwyn, G. *et al.* International Patient Decision Aids Standards (IPDAS) Collaboration. Developing a quality criteria framework for patient decision aid: online international Delphi consensus process. *Br. Med. J.* **333**, 417–419 (2006).
- 72. Schapira, M. M. et al. The Impact of a Risk-Based Breast Cancer Screening Decision Aid on Initiation of Mammography Among Younger Women: Report of a Randomized Trial. *MDM Policy Pract.* **4**, 2381468318812889 (2019).
- 73. Seitz, H. H. *et al.* Explaining the effects of a decision intervention on mammography intentions: The roles of worry, fear and perceived susceptibility to breast cancer. *Psychol. Health* **33**, 682–700 (2018).
- 74. Bonner, C. *et al.* I Don't Believe It, But I'd Better Do Something About It: Patient Experiences of Online Heart Age Risk Calculators. *J. Med. Internet Res.* **16**, e120 (2014).
- 75. McCaffery, K. *et al.* How different terminology for ductal carcinoma in situ impacts women's concern and treatment preferences: a randomised comparison within a national community survey. *BMJ Open* **5**, e008094 (2015).
- 76. Nickel, B., Barratt, A., Copp, T., Moynihan, R. & McCaffery, K. Words do matter: a systematic review on how different terminology for the same condition influences management preferences. *BMJ Open* **7**, e014129 (2017).
- 77. Brandhof, S. D. *et al.* Colorectal cancer screening: Associations between information provision, attitudes and intended participation. *Patient Educ. Couns.* **101**, 546–550 (2018).
- 78. Copp, T. *et al.* Influence of the disease label 'polycystic ovary syndrome' on intention to have an ultrasound and psychosocial outcomes: a randomised online study in young women. *Hum. Reprod.* **32**, 876–884 (2017).
- 79. Hersch, J., Jansen, J. & McCaffery, K. Decision-making about mammographic screening: pursuing informed choice. *Climacteric* **21**, 209–213 (2018).
- 80. Hersch, J. *et al.* Overdetection in breast cancer screening: development and preliminary evaluation of a decision aid. *BMJ Open 4*, e006016–e006016 (2014).
- 81. Lewis, C. L., Brenner, A. T., Griffith, J. M. & Pignone, M. P. The uptake and effect of a mailed multi-modal colon cancer screening intervention: A pilot controlled trial. *Implement. Sci.* **3**, 32 (2008).
- 82. Griffith, J. M., Lewis, C. L., Brenner, A. R. & Pignone, M. P. The effect of offering different numbers of colorectal cancer screening test options in a decision aid: a pilot randomized trial. *BMC Med. Inform. Decis. Mak.* **8**, 4 (2008).
- 83. Kim, J. *et al.* Development and initial testing of a computer-based patient decision aid to promote colorectal cancer screening for primary care practice. *BMC Med. Inform. Decis. Mak.* **5**, 36 (2005).
- 84. Fagerlin, A., Zikmund-Fisher, B. J. & Ubel, P. A. Helping Patients Decide: Ten Steps to Better Risk Communication. *J. Natl. Cancer Inst.* **103**, 1436–1443 (2011).
- 85. Lewis, C. L. *et al.* Older adults' attitudes about continuing cancer screening later in life: a pilot study interviewing residents of two continuing care communities. *BMC Geriatr.* **6**, 10 (2006).
- 86. Piper, M. S. *et al.* Patient Attitudes Toward Individualized Recommendations to Stop Low-Value Colorectal Cancer Screening. *JAMA Netw. Open* **1**, e185461–e185461 (2018).
- 87. Dillard, A. J. *et al.* Breast cancer anxiety's associations with responses to a chemoprevention decision aid. *Soc. Sci. Med.* **77**, 13–19 (2013).

- 88. Dillard, A. J., Scherer, L. D., Ubel, P. A., Alexander, S. & Fagerlin, A. Anxiety symptoms prior to a prostate cancer diagnosis: Associations with knowledge and openness to treatment. *Br. J. Health Psychol.* **22**, 151–168 (2017).
- 89. Hoerger, M., Scherer, L. D. & Fagerlin, A. Affective Forecasting and Medication Decision Making in Breast Cancer Prevention. *Health Psychol. Off. J. Div. Health Psychol. Am. Psychol. Assoc.* **35**, 594–603 (2016).
- 90. Kang, S. K. *et al.* A Randomized Study of Patient Risk Perception for Incidental Renal Findings on Diagnostic Imaging Tests. *Am. J. Roentgenol.* **210**, 369–375 (2018).
- 91. Rothberg, M. B. *et al.* The Effect of Information Presentation on Beliefs About the Benefits of Elective Percutaneous Coronary Intervention. *JAMA Intern. Med.* **174**, 1623–1629 (2014).
- 92. Breast Cancer Risk Assessment Tool. *Breast Cancer Risk Assessment Tool* https://www.cancer.gov/bcrisktool.
- 93. Housten, A. J. *et al.* A Review of the Presentation of Overdiagnosis in Cancer Screening Patient Decision Aids. *MDM Policy Pract.* **4**, 2381468319881447 (2019).
- 94. Anderson, L. R. Belief defense produced by derogation of message source. *J. Exp. Soc. Psychol.* **3**, 349–360 (1967).
- 95. Zhao, X., Strasser, A., Cappella, J. N., Lerman, C. & Fishbein, M. A measure of perceived argument strength: Reliability and validity. *Commun. Methods Meas.* **5**, 48–75 (2011).
- 96. Egede, L. E. & Ellis, C. Development and Testing of the Multidimensional Trust in Health Care Systems Scale. *J. Gen. Intern. Med.* **23**, 808–815 (2008).
- 97. Fagerlin, A. *et al.* Measuring numeracy without a math test: Development of the subjective numeracy scale. *Med. Decis. Making* **27**, 672–680 (2007).
- 98. Chew, L. D. *et al.* Validation of Screening Questions for Limited Health Literacy in a Large VA Outpatient Population. *J. Gen. Intern. Med.* **23**, 561–566 (2008).
- 99. Petrova, D., Garcia-Retamero, R. & Cokely, E. T. Understanding the Harms and Benefits of Cancer Screening: A Model of Factors That Shape Informed Decision Making. *Med. Decis. Making* **35**, 847–858 (2015).